CLINICAL TRIAL: NCT00135824
Title: Local Tolerability and Safety of Povidone K25 (Artificial Tears Containing Povidone) vs. Placebo in Healthy Volunteers
Brief Title: Local Tolerability and Safety of Povidone K25 Eye Drops (Artificial Tears Containing Povidone) Versus Placebo in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COCF355ADE01
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-11

CONDITIONS: Healthy
Keywords: Artificial eye drops; tolerability; healthy volunteers; povidone; healthy subjects
MeSH Terms: interventions — Povidone

INTERVENTIONS:
Drug: Povidone K25 eye drops (povidone)

SUMMARY:
Instillation of artificial tears is standard treatment in dry eye syndrome and in patients experiencing dry eye symptoms when wearing contact lenses. Povidone K25 eye drops (povidone) is an isotonic solution containing povidone to simulate normal tears viscosity. Safety and local tolerability of Povidone K25 is evaluated in healthy volunteers in comparison to placebo eye drops.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Older than 18 years
* Ocular discomfort less than 20 mm on 100 mm visual analogue scale (VAS) prior to treatment

Exclusion Criteria:

* Known hypersensitivity to any of the constituents of the medications
* Known allergic disposition (e.g. hay fever)
* Wearing of contact lenses
* Any kind of current eye disease (e.g. dry eye)

Additional exclusion criteria are defined in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-03; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
ocular discomfort by using a visual analogue scale (VAS)

SECONDARY OUTCOMES:
slit lamp assessment (conjunctival edema, palpebral hyperemia, lid edema)
adverse events

CONTACTS AND LOCATIONS:
Overall Officials: PD. Dr. G. Auffarth, Principal Investigator — Universitäts-Augenklinik, Im Neuenheimer Feld 400,
Locations (1):
- Novartis Investigational Site, Heidelberg, Germany